CLINICAL TRIAL: NCT02157480
Title: ELECTRODIAB2: Effect of an Outpatient Program of Bi-quadricipital Electrostimulation on Glucose Profile of Sedentary Patients With Type 2 Diabetes.
Brief Title: Effect of Electrostimulation on Glucose Profile of Patients With Type 2 Diabetes
Acronym: ELECTRODIAB2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: University Hospital, Rouen (Other); Amiens University Hospital (Other); University Hospital, Lille (Other); General Hospital Roubaix (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00231-46
Record Dates: First submitted 2014-05-19; First posted 2014-06-06 (Estimated); Last update posted 2022-08-24 (Actual); Status verified 2022-07

CONDITIONS: Type 2 Diabetes; Physical Activity
Keywords: glucose profile; continuous glucose monitoring; electrostimulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (No Intervention): usual follow-up for 6 weeks
- electrostimulation 3 days per week (Experimental): 20 minutes ambulatory bi-quadricipital electrostimulation sessions three times per week for 6 weeks
  Interventions: Device: electrostimulation (with Compex® Compex2* (DJO, Vista, CA, USA)) 3 days per week .
- electrostimulation 5 days per week (Experimental): 20 minutes ambulatory bi-quadricipital electrostimulation sessions five times per week for 6 weeks
  Interventions: Device: electrostimulation (with Compex® Compex2* (DJO, Vista, CA, USA)) 5 days per week

INTERVENTIONS:
Device: electrostimulation (with Compex® Compex2* (DJO, Vista, CA, USA)) 3 days per week . — outpatient biquadricipital electrostimulation 3 days per week with an electrostimulator Compex2* (DJO, Vista, CA, USA)
  Arms: electrostimulation 3 days per week
Device: electrostimulation (with Compex® Compex2* (DJO, Vista, CA, USA)) 5 days per week — outpatient biquadricipital electrostimulation 5 days per week with an electrostimulator Compex2* (DJO, Vista, CA, USA)
  Arms: electrostimulation 5 days per week

SUMMARY:
Prevalence of type 2 diabetes (T2D) is increasing worldwide. Lifestyle remains the cornerstone treatment for patients with T2D who are often overweight and sedentary.

Physical activity improves glucose metabolism of patients with T2D : increased glucose utilization during acute muscle activity and improved insulin sensitivity after regular training. The molecular mechanism underlying the effects of exercise on glucose metabolism involves the glucose transporter GLUT-4 which is regulated by physical activity.

Several studies and meta-analysis have showed that physical activity reduces HbA1c by 0.6% on average. In addition, other data suggest a decrease in cardiovascular morbidity and mortality through physical activity.

Recent recommendations for T2D management call for the practice of a structured type of endurance 150 minutes per week and muscle building 2 times per week. However, implementation of these recommendations is low, even when integrated into a therapeutic education program. Adherence is often transient and / or partial. In addition, many T2D subjects are unable to initiate a physical activity because of disabling complications or comorbidities or because of a major cardiorespiratory deconditioning.

Neuro-myo electrical stimulation (NMES) is a physical treatment routinely used in functional rehabilitation to improve muscle strength and volume. The metabolic effect of NMES has been little studied. A pilot study conducted by our team on a population of 18 subjects with T2D showed that a week of daily NMES sessions significantly improved insulin sensitivity of about 25% and up to 50 % for good responders. This result contrasted with the low induced energy expenditure by each 20-minute session of bi-quadricipital NMES, suggesting the possibility of a humoral or neural mechanism associated with NMES.

To complete this work, we plan a randomized cross-over trial with 3 periods (6 weeks without NMES (control), 6 weeks with 3 sessions of NMES per week and 6 weeks with 5 sessions of NMES per week) to assess the glucose profile of sedentary T2D subjects during these different periods. We hypothesize that the bi-quadricipital NMES could improve glycemic control in T2D subjects and thus represent an alternative to traditional physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes treated with lifestyle, oral hypoglycemic agents and/or GLP-1 agonists.
* HbA1c : 7 to 10%
* low physical activity (Ricci and Gagnon score below 27)
* Insulin-resistance (at least one criteria out three):
* Waist circumference > 80cm in women and > 94cm in men
* Triglycerides > 150 mg/dl
* HDL-c < 50 mg/dl for women, < 40 mg/dl for men

Exclusion Criteria:

* type 1 diabetes
* pregnancy
* intense usual physical activity
* pace maker
* seizure
* knee or neuromuscular pathology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-09; Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Mean CGM glucose from a 6-day CGM recording | week 0, 6, 13, 20

SECONDARY OUTCOMES:
HbA1c | week 0, 6, 13, 20

OTHER OUTCOMES:
fasting plasma glucose | Week 0, 6, 13, 20
fasting plasma insulin | Week 0, 6, 13, 20
FFA (free fatty acid) | Week 0, 6, 13, 20
IL6 (interleukin 6) | Week 0, 6, 13, 20
TNFalpha | Week 0, 6, 13, 20
adiponectin | Week 0, 6, 13, 20
CRPus (C Reactive Protein ultra sensitive) | Week 0, 6, 13, 20
irisin | Week 0, 6, 13, 20
satisfaction questionnaire | Week 0, 6, 13, 20
motivation questionnaire for physical activity | Week 0, 6, 13, 20
cardiometabolic stress test | Week 6, 20

CONTACTS AND LOCATIONS:
Overall Officials: Corinne FOURMY, MD, Principal Investigator — University Hospital, Caen
Locations (5):
- France (5):
  - University Hospital Amiens, Amiens
  - Clinical Research Center University Hospital Caen, Caen
  - University Hospital Lille, Lille
  - General Hospital Roubaix, Roubaix
  - CHU Rouen, Rouen